CLINICAL TRIAL: NCT03795714
Title: Intravascular Ultrasound and Optical Coherence Tomography-Defined Optimal Criteria and Plaque Characteristics for Defining the Functional Significance of Coronary Stenoses Using Resting and Hyperemic Physiologic Indices
Brief Title: Association Between IVUS and OCT Parameters and Invasive Physiologic Indices
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: IVUS2017-11-056-001
Record Dates: First submitted 2018-12-28; First posted 2019-01-08 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Ischemic Heart Disease
Keywords: Intravascular Ultrasound; Optical Coherence Tomography; Fractional Flow Reserve; Diastolic Pressure Ratio; Resting Full-Cycle Ratio; Ischemic Heart Disease; Instantaneous Wave-free Ratio
MeSH Terms: conditions — Myocardial Ischemia | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intravascular Imaging and Physiologic Assessment: 330 patients with suspected ischemic heart disease and who underwent IVUS or OCT assessment and invasive physiologic assessment.
  Interventions: Diagnostic Test: IVUS or OCT and Invasive physiologic indices

INTERVENTIONS:
Diagnostic Test: IVUS or OCT and Invasive physiologic indices — IVUS or OCT measurement in order to evaluate the lesion morphology and stent optimization, and invasive physiologic measurement in order to functional significance of epicardial stenosis

SUMMARY:
1. to evaluate diagnostic accuracy and performance of IVUS and OCT-derived quantitative parameters to predict functional significance of stenosis defined using all the available physiologic indices.
2. to explores the association between intravascular imaging-derived plaque characteristics and invasive physiologic indices.

DETAILED DESCRIPTION:
Given the inherent limitations of coronary angiography to depict the presence of functionally significant epicardial coronary stenosis and discrepancy between angiographic stenosis severity and the presence of myocardial ischemia, invasive physiologic indices such as fractional flow reserve (FFR) or instantaneous wave-free ratio (iFR) has been a standard method to guide decision of revascularization.

Intravascular ultrasound (IVUS) and optical coherence tomography (OCT) are an intracoronary imaging method able to provide information about lumen area, vessel area, plaque burden, and plaque characteristics that can be used for the guidance of revascularization procedure. Several previous studies explored the diagnostic performance of intravascular imaging-defined quantitative parameters to predict functional significance defined by FFR, however, quantitative parameter derived from intravascular imaging showed only moderate diagnostic accuracy and the optimal cut-off value of intravascular imaging-derived minimal lumen area (MLA) or minimal lumen diameter (MLD) were varied according to the patient population, interrogated vessels, and the location of target lesions, suggesting limited clinical relevance of judging functional significance of target stenosis using intravascular imaging alone. Nevertheless, the adoption rate of FFR-guided decision has been limited due to various reasons and intravascular image-guided decision has been still used in substantial proportion of the patients.

Recently, new resting pressure-derived indices including resting full-cycle ratio (RFR) or diastolic pressure ratio (dPR) have been introduced as other substitutes for iFR, which does not require administration of hyperemic agents, therefore, possess more convenient in daily practice. Recent study with the largest sample size demonstrated identical diagnostic property and prognostic implication among iFR, RFR, and dPR. As those resting pressure-derived indices might have more generalizability for daily practice, it is expected to raise the adoption rate of physiologic interrogation. Therefore, understanding the association between all the available physiologic indices and intravascular imaging-derived quantitative and qualitative parameters might be important in clinical decision for patient who underwent invasive coronary angiography.

In this regard, the investigators sought to evaluate diagnostic accuracy and performance of intravascular imaging-derived quantitative parameters to predict functional significance of stenosis defined using all the available physiologic indices and further explores the association between IVUS and OCT-derived plaque characteristics and invasive physiologic indices.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suspected ischemic heart disease, and underwent invasive physiologic assessment and intravascular ultrasound

Exclusion Criteria:

* Cardiogenic shock
* Graft vessel
* In-stent restenosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 330 patients with suspected ischemic heart disease and who underwent IVUS or OCT assessment and invasive physiologic assessment.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by fractional flow reserve (FFR) | During Cardiac Cath
  Diagnostic accuracy of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Diagnostic accuracy of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by instantaneous wave-free ratio (iFR) | During Cardiac Cath
  Diagnostic accuracy of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Diagnostic accuracy of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by diastolic pressure ratio (dPR) | During Cardiac Cath
  Diagnostic accuracy of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Diagnostic accuracy of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by resting full-cycle ratio (RFR) | During Cardiac Cath
  Diagnostic accuracy of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Diagnostic accuracy of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Diagnostic accuracy of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Diagnostic accuracy of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Diagnostic accuracy of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Diagnostic accuracy of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Diagnostic accuracy of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Diagnostic accuracy of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Diagnostic accuracy of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Diagnostic accuracy of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Diagnostic accuracy of minimal lumen area assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Diagnostic accuracy of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Diagnostic accuracy of minimal lumen area assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Diagnostic accuracy of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Diagnostic accuracy of minimal lumen area assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Diagnostic accuracy of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Diagnostic accuracy of minimal lumen area assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Diagnostic accuracy of plaque burden assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Diagnostic accuracy of plaque burden assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Diagnostic accuracy of plaque burden assessed by IVUS to predict functional significance assessed by iFR | During Cardiac Cath
  Diagnostic accuracy of plaque burden assessed by IVUS to predict functional significance defined by iFR ≤0.89
Diagnostic accuracy of plaque burden assessed by IVUS to predict functional significance assessed by dPR | During Cardiac Cath
  Diagnostic accuracy of plaque burden assessed by IVUS to predict functional significance defined by dPR ≤0.89
Diagnostic accuracy of plaque burden assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Diagnostic accuracy of plaque burden assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89

SECONDARY OUTCOMES:
Sensitivity of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Sensitivity of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Sensitivity of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Sensitivity of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Sensitivity of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Sensitivity of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Sensitivity of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Sensitivity of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Sensitivity of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Sensitivity of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Sensitivity of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Sensitivity of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Sensitivity of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Sensitivity of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Sensitivity of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Sensitivity of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Sensitivity of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Sensitivity of minimal lumen area assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Sensitivity of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Sensitivity of minimal lumen area assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Sensitivity of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Sensitivity of minimal lumen area assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Sensitivity of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Sensitivity of minimal lumen area assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Sensitivity of plaque burden assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Sensitivity of plaque burden assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Sensitivity of plaque burden assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Sensitivity of plaque burden assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Sensitivity of plaque burden assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Sensitivity of plaque burden assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Sensitivity of plaque burden assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Sensitivity of minimal lumen area assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Specificity of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Specificity of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Specificity of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Specificity of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Specificity of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Specificity of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Specificity of percent diameter stenosis assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Specificity of percent diameter stenosis assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Specificity of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Specificity of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Specificity of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Specificity of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Specificity of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Specificity of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Specificity of minimal lumen diameter assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Specificity of minimal lumen diameter assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Specificity of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Specificity of minimal lumen area assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Specificity of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Specificity of minimal lumen area assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Specificity of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Specificity of minimal lumen area assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Specificity of minimal lumen area assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Specificity of minimal lumen area assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Specificity of plaque burden assessed by intravascular imaging to predict functional significance assessed by FFR | During Cardiac Cath
  Specificity of plaque burden assessed by intravascular imaging to predict functional significance defined by FFR ≤0.80
Specificity of plaque burden assessed by intravascular imaging to predict functional significance assessed by iFR | During Cardiac Cath
  Specificity of plaque burden assessed by intravascular imaging to predict functional significance defined by iFR ≤0.89
Specificity of plaque burden assessed by intravascular imaging to predict functional significance assessed by dPR | During Cardiac Cath
  Specificity of plaque burden assessed by intravascular imaging to predict functional significance defined by dPR ≤0.89
Specificity of plaque burden assessed by intravascular imaging to predict functional significance assessed by RFR | During Cardiac Cath
  Specificity of plaque burden assessed by intravascular imaging to predict functional significance defined by RFR ≤0.89
Linear correlation between percent diameter stenosis and FFR | During Cardiac Cath
  Linear regression analysis between percent diameter stenosis and FFR
Linear correlation between percent diameter stenosis and iFR | During Cardiac Cath
  Linear regression analysis between percent diameter stenosis and iFR
Linear correlation between percent diameter stenosis and dPR | During Cardiac Cath
  Linear regression analysis between percent diameter stenosis and dPR
Linear correlation between percent diameter stenosis and RFR | During Cardiac Cath
  Linear regression analysis between percent diameter stenosis and RFR
Linear correlation between minimal lumen diameter and FFR | During Cardiac Cath
  Linear regression analysis between minimal lumen diameter and FFR
Linear correlation between minimal lumen diameter and iFR | During Cardiac Cath
  Linear regression analysis between minimal lumen diameter and iFR
Linear correlation between minimal lumen diameter and dPR | During Cardiac Cath
  Linear regression analysis between minimal lumen diameter and dPR
Linear correlation between minimal lumen diameter and RFR | During Cardiac Cath
  Linear regression analysis between minimal lumen diameter and RFR
Linear correlation between minimal lumen area and FFR | During Cardiac Cath
  Linear regression analysis between minimal lumen area and FFR
Linear correlation between minimal lumen area and iFR | During Cardiac Cath
  Linear regression analysis between minimal lumen area and iFR
Linear correlation between minimal lumen area and dPR | During Cardiac Cath
  Linear regression analysis between minimal lumen area and dPR
Linear correlation between minimal lumen area and RFR | During Cardiac Cath
  Linear regression analysis between minimal lumen area and RFR
Linear correlation between plaque burden and FFR | During Cardiac Cath
  Linear regression analysis between plaque burden and FFR
Linear correlation between plaque burden and iFR | During Cardiac Cath
  Linear regression analysis between plaque burden and iFR
Linear correlation between plaque burden and dPR | During Cardiac Cath
  Linear regression analysis between plaque burden and dPR
Linear correlation between plaque burden and RFR | During Cardiac Cath
  Linear regression analysis between plaque burden and RFR
Discriminatory function of percent diameter stenosis to predict functional significance assessed by FFR | During Cardiac Cath
  Discriminatory function of percent diameter stenosis to predict functional significance defined by FFR≤0.80
Discriminatory function of percent diameter stenosis to predict functional significance assessed by iFR | During Cardiac Cath
  Discriminatory function of percent diameter stenosis to predict functional significance defined by iFR≤0.89
Discriminatory function of percent diameter stenosis to predict functional significance assessed by dPR | During Cardiac Cath
  Discriminatory function of percent diameter stenosis to predict functional significance defined by dPR≤0.89
Discriminatory function of percent diameter stenosis to predict functional significance assessed by RFR | During Cardiac Cath
  Discriminatory function of percent diameter stenosis to predict functional significance defined by RFR≤0.89
Discriminatory function of minimal lumen diameter to predict functional significance assessed by FFR | During Cardiac Cath
  Discriminatory function of minimal lumen diameter to predict functional significance defined by FFR≤0.80
Discriminatory function of minimal lumen diameter to predict functional significance assessed by iFR | During Cardiac Cath
  Discriminatory function of minimal lumen diameter to predict functional significance defined by iFR≤0.89
Discriminatory function of minimal lumen diameter to predict functional significance assessed by dPR | During Cardiac Cath
  Discriminatory function of minimal lumen diameter to predict functional significance defined by dPR≤0.89
Discriminatory function of minimal lumen diameter to predict functional significance assessed by RFR | During Cardiac Cath
  Discriminatory function of minimal lumen diameter to predict functional significance defined by RFR≤0.89
Discriminatory function of minimal lumen area to predict functional significance assessed by FFR | During Cardiac Cath
  Discriminatory function of minimal lumen area to predict functional significance defined by FFR≤0.80
Discriminatory function of minimal lumen area to predict functional significance assessed by iFR | During Cardiac Cath
  Discriminatory function of minimal lumen area to predict functional significance defined by iFR≤0.89
Discriminatory function of minimal lumen area to predict functional significance assessed by dPR | During Cardiac Cath
  Discriminatory function of minimal lumen area to predict functional significance defined by dPR≤0.89
Discriminatory function of minimal lumen area to predict functional significance assessed by RFR | During Cardiac Cath
  Discriminatory function of minimal lumen area to predict functional significance defined by RFR≤0.89
Discriminatory function of plaque burden to predict functional significance assessed by FFR | During Cardiac Cath
  Discriminatory function of plaque burden to predict functional significance defined by FFR≤0.80
Discriminatory function of plaque burden to predict functional significance assessed by iFR | During Cardiac Cath
  Discriminatory function of plaque burden to predict functional significance defined by iFR≤0.89
Discriminatory function of plaque burden to predict functional significance assessed by dPR | During Cardiac Cath
  Discriminatory function of plaque burden to predict functional significance defined by dPR≤0.89
Discriminatory function of plaque burden to predict functional significance assessed by RFR | During Cardiac Cath
  Discriminatory function of plaque burden to predict functional significance defined by RFR≤0.89

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Study Chair — Professor; Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Assistant Professor
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul national university hospital, Seoul

REFERENCES:
- [Derived] Lee JM, Choi KH, Koo BK, Zhang J, Han JK, Yang HM, Park KW, Song YB, Hahn JY, Choi SH, Gwon HC, Kim HS. Intravascular ultrasound or optical coherence tomography-defined anatomic severity and hemodynamic severity assessed by coronary physiologic indices. Rev Esp Cardiol (Engl Ed). 2020 Oct;73(10):812-821. doi: 10.1016/j.rec.2019.11.001. Epub 2019 Dec 4. English, Spanish. PMID 31812517